CLINICAL TRIAL: NCT05130242
Title: Posterior Instrumentation for Osteoporotic Fractures in the Thoracic or Lumbar Spine: A Retrospective Comparison Between Cement Augmented Pedicle Screws and Hybrid Constructs of Pedicle Screws and Hooks
Brief Title: A Retrospective Comparison Between CPS and HC Techniques for Osteoporotic Fractures in the Thoracic or Lumbar Spine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-01-030CC
Record Dates: First submitted 2021-10-19; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Osteoporosis
Keywords: Thoracolumbar fracture; Cement augmentation; Hook; Pedicle Screw; Hybrid Construct
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cement-augmented Pedicle Screws (CPS) Group
  Interventions: Procedure: Cement-augmented Pedicle Screws (CPS)
- Hybrid Construct (HC) group
  Interventions: Procedure: Hybrid Construct (HC)

INTERVENTIONS:
Procedure: Cement-augmented Pedicle Screws (CPS) — Patients who received surgical treatment with CPS for osteoporotic fractures in the thoracic or lumbar spine
  Groups: Cement-augmented Pedicle Screws (CPS) Group
Procedure: Hybrid Construct (HC) — Patients who received surgical treatment with HC consisting of pedicle screws and additional hooks for osteoporotic fractures in the thoracic or lumbar spine
  Groups: Hybrid Construct (HC) group

SUMMARY:
Cement-augmented pedicle screws (CPS) and hybrid construct (HC) consisting of pedicle screws and additional hooks are common methods in osteoporotic fracture of the thoracic and lumbar spine. No study has compared the surgical results between CPS and HC techniques for treatment of the osteoporotic thoracic and lumbar spine fracture. The aim of the retrospective study was to compare surgical results using CPS or HC for osteoporotic fractures in the thoracic or lumbar spine. Patients who received surgical treatment with CPS or HC for osteoporotic fractures in the thoracic or lumbar spine.

DETAILED DESCRIPTION:
Osteoporosis, the most common metabolic bone disease, leads to alteration of bone density that has been shown to compromise the strength of spinal instrumentation. With elderly populations growing, rates of spine surgery performed on osteoporotic patients have increased to treat a variety of conditions. Vertebral fracture is the most common osteoporotic fracture in the elderly, and surgical intervention is sometimes needed for patients who are diagnosed as nonunion, failure of vertebroplasty, and neurologic deficits. Therefore, spine surgeons will increasingly face the challenge of achieving rigid fixation of osteoporotic spines.

Cement-augmented pedicle screws are the most common strategy to maximize pullout strength for fixation of osteoporotic spines. Hybrid constructs, a combination of pedicle screws and hooks, offer an alternative approach to avoid implant failure and increasing construct stability when placing instrumentation in the osteoporotic spine. Biomechanical studies of either cement-augmented pedicle screws or combined pedicle screws and hooks for osteoporotic spine have demonstrated superior results compared to pedicle screws only in terms of improving implant pullout strength. However, few clinical investigation to date has focused on comparing surgical results of the cement-augmented pedicle screws (CPS) and hybrid construct (HC) techniques. The goal of the retrospective cohort study was to compare the surgical outcomes and surgery-, patient- and implant-related complications between the CPS and HC techniques for osteoporotic vertebral fractures in the thoracic or lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* Surgical treatment with CPS or HC of pedicle screws and hooks for osteoporotic fractures in the thoracic or lumbar spine
* Received a minimum of 2-year follow-up

Exclusion Criteria:

* T-scores greater than -2.5
* Cancer metastasis
* Chronic osteomyelitis
* Failure to complete the questionnaires or radiographic examinations

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent surgical treatment with CPS or HC of pedicle screws and hooks for osteoporotic fractures in the thoracic or lumbar spine in our hospital from January 2011 through December 2015
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-01-21 (Estimated); Study Completion 2022-01-21 (Estimated)

PRIMARY OUTCOMES:
Implant Failure | Postoperative 1 year
  Implant failure was defined as pull-out or breakage of the implants on plain X-ray film.
Kyphotic Angle | Preoperative
  Cobb's method was used to measure the regional kyphotic angle
Kyphotic Angle | Postoperative 1 month.
  Cobb's method was used to measure the regional kyphotic angle
Kyphotic Angle | Postoperative 2 months.
  Cobb's method was used to measure the regional kyphotic angle
Kyphotic Angle | Postoperative 3 months.
  Cobb's method was used to measure the regional kyphotic angle
Kyphotic Angle | Postoperative 6 months.
  Cobb's method was used to measure the regional kyphotic angle
Kyphotic Angle | Postoperative 12 months.
  Cobb's method was used to measure the regional kyphotic angle
Visual Analogue Scale (VAS) | Preoperative
  Functional outcomes, Back pain evaluated
Visual Analogue Scale (VAS) | Postoperative 1 month.
  Functional outcomes, Back pain evaluated
Visual Analogue Scale (VAS) | Postoperative 2 months.
  Functional outcomes, Back pain evaluated
Visual Analogue Scale (VAS) | Postoperative 3 months.
  Functional outcomes, Back pain evaluated
Visual Analogue Scale (VAS) | Postoperative 6 months.
  Functional outcomes, Back pain evaluated
Visual Analogue Scale (VAS) | Postoperative 12 months.
  Functional outcomes, Back pain evaluated
Oswestry Disability Index (ODI) | Preoperative
  Functional outcomes, Disability evaluated
Oswestry Disability Index (ODI) | Postoperative 1 month.
  Functional outcomes, Disability evaluated
Oswestry Disability Index (ODI) | Postoperative 2 months.
  Functional outcomes, Disability evaluated
Oswestry Disability Index (ODI) | Postoperative 3 months.
  Functional outcomes, Disability evaluated
Oswestry Disability Index (ODI) | Postoperative 6 months.
  Functional outcomes, Disability evaluated
Oswestry Disability Index (ODI) | Postoperative 12 months.
  Functional outcomes, Disability evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Orthopedics and Traumatology, Taipei Veterans General Hospital, Taipei, Taiwan